CLINICAL TRIAL: NCT04237753
Title: Optimizing Remote Access to Urinary Incontinence Treatment for Women Veterans
Brief Title: Remote Access to Urinary Incontinence Treatment for Women Veterans
Acronym: PRACTICAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IIR 18-266
Record Dates: First submitted 2019-12-31; First posted 2020-01-23 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Urinary Incontinence
Keywords: women's health; Veterans; telemedicine; urinary incontinence; overactive urinary bladder; urinary bladder diseases; stress urinary incontinence; urge urinary incontinence; health education
MeSH Terms: conditions — Urinary Incontinence; Urinary Bladder, Overactive; Urinary Bladder Diseases; Urinary Incontinence, Stress; Urinary Incontinence, Urge; Health Education

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial with adaptive trial design. Randomization will first involve treatment with one of two delivery methods: (1) a web-based mobile health application or (2) a single video session. For women who do not improve (SMART design), they will receive a first or second video session.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MyHealthebladder (Active Comparator): Daily mobile health education with information on bladder anatomy and function, pelvic floor muscle exercises with behavioral strategies, and self-monitoring tools for urine leakage
  Interventions: Behavioral: MyHealtheBladder
- VA Video Connect (Active Comparator): Remote telehealth visits with continence care provider who will provide education on bladder anatomy and function, pelvic floor muscle exercises with behavioral strategies, and self-monitoring tools for urine leakage
  Interventions: Behavioral: VA Video Connect

INTERVENTIONS:
Behavioral: VA Video Connect — Remote telehealth visits with continence care provider who will provide education on bladder anatomy and function, pelvic floor muscle exercises with behavioral strategies, and self-monitoring tools for urine leakage
  Other Names: Telehealth visit with Continence Provider
  Arms: VA Video Connect
Behavioral: MyHealtheBladder — Daily mobile health education with information on bladder anatomy and function, pelvic floor muscle exercises with behavioral strategies, and self-monitoring tools for urine leakage
  Other Names: Mobile health bladder education
  Arms: MyHealthebladder

SUMMARY:
This study is about assessing the helpfulness of two treatment delivery methods for bladder leakage or urinary incontinence. It is being funded by the Department of Veterans Affairs. By doing this study, the investigators hope to learn which treatment method is the most helpful remote delivery method for treating bladder leakage. The total participation time in this research is 6 months. During the first 8 -12 weeks of the study, you will receive standard of care from an online educational program (MyHealtheBladder) or a video visit with a provider through VA Video Connect. You will be selected by chance to receive MyHealtheBladder or VA Video Connect. About half-way through the study, the investigators will ask you about your bladder symptoms. If your bladder symptoms are not better, you will be selected by chance to continue the previous treatment or receive an initial or booster video session with a provider. Throughout the study, you will be asked to answer questions related to your health, bladder leakage, costs due to bladder leakage, and track your behavioral training.

DETAILED DESCRIPTION:
This study represents a unique opportunity to improve access to treatments for urine leakage for women Veterans. This research study will examine the effects of two mobile health technologies on improving bladder symptoms, as part of a randomized clinical trial. The study includes 260 women Veterans recruited from 3 sites: the Birmingham VAMC, the Atlanta VAHCS, and the Durham VAMC (86 per site). Women will receive first-line treatments for urine leakage through randomization to one of two delivery methods for direct treatment: (1) a web-based mobile health application that delivers content daily for 8 weeks compared to (2) a single video session delivered by VA Video Connect. At 8-weeks, women who do not have improved symptoms will have the ability to continue the treatment or receive an initial or booster video session. The investigators will measure bladder symptoms (3 questions by self-report over the phone or via survey) at baseline, 8-weeks, 12-weeks, and 6-months. Additionally, the investigators will interview 54 women Veterans and 12 providers to learn about their experiences with the technologies using 1:1 telephone interviews at 12-weeks. The findings from this study will inform the best technology to improve access for bladder leakage among women Veterans across a wider array of VHA facilities.

ELIGIBILITY:
Inclusion Criteria:

* Women Veterans
* Urinary incontinence occurring at least monthly for 3 months
* Able to access daily internet via computer or mobile device
* Access to personal email for MyHealtheBladder and VA Video Connect visit initiation and reminder

Exclusion Criteria:

* Unstable medical conditions that could contribute to incontinence (e.g., recent major hospitalization, planned major surgery, conditions that affect urine volume - hemoglobin A1c of 9.0, chronic kidney disease with planned dialysis within 3 months, as assessed by PI or Site PI)
* Unstable psychiatric conditions (e.g., psychosis, suicidal, active alcohol/substance abuse based on history and medical records)
* Unstable housing situation
* Genitourinary cancer undergoing active treatment with chemotherapy or radiation
* Neurologic conditions known to contribute to incontinence (Multiple Sclerosis, Parkinson's Disease, TBI, Dementia, and Stroke Survivors with limited mobility)
* New treatments for incontinence started in the prior 3 months or planned during the 6-month study duration, includes medications and/or surgery
* Three months post-partum

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 286 (Actual)
Dates: Start 2020-04-06 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Change in International Consultation on Incontinence Questionnaire - Urinary Incontinence Short Form (ICIQ-UI SF) | baseline to 12 weeks
  Urinary incontinence severity questionnaire, range 0-21, higher scores represent greater symptom severity

SECONDARY OUTCOMES:
Change International Consultation on Incontinence Modular Questionnaire (ICIQ)-Overactive Bladder (OAB) | baseline to 12-weeks
  Overactive bladder symptom severity questionnaire, range 0-12, higher scores represent greater symptoms severity
Global Rating of Patient Satisfaction | 12-weeks
  Patient satisfaction question (PSQ) - 3 categories of response (highly satisfied, satisfied, not satisfied)
Self-reported Pelvic floor muscle exercise adherence | 12-weeks
  Adherence to pelvic floor muscle exercises reported as exercises per day completed over each week. Adherence defined as 80% of days with exercises completed over 12-week intervention period.
Change in International Consultation on Incontinence Modular Questionnaire (ICIQ)- Urinary Incontinence Short Form (ICIQ-UI SF) | baseline to 24-weeks
  Urinary incontinence severity questionnaire, range 0-21, higher scores represent greater symptom severity, longer term outcome

OTHER OUTCOMES:
Miles saved | 12-weeks
  Mean miles saved from home location to specialty care clinic location over 12-week intervention

CONTACTS AND LOCATIONS:
Overall Officials: Alayne D Markland, DO MSc, Principal Investigator — Birmingham VA Medical Center, Birmingham, AL; Elizabeth Camille Vaughan, MD MS, Principal Investigator — Atlanta VA Medical and Rehab Center, Decatur, GA; Susan N. Hastings, MD MHSc, Principal Investigator — Durham VA Medical Center, Durham, NC
Locations (3):
- United States (3):
  - Birmingham VA Medical Center, Birmingham, AL, Birmingham, Alabama
  - Atlanta VA Medical and Rehab Center, Decatur, GA, Decatur, Georgia
  - Durham VA Medical Center, Durham, NC, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: Yes
For purposes of this study, all data will be stripped of all patient identifiers and each participant will be given a unique identifier for the study. Participant records will be stored in a locked cabinet in a locked office and will be accessible only to the Principal Investigator, Nurse Practitioner delivering the intervention, Research Coordinator, and Site PI's (Markland, Vaughan, and Goldstein) and co-investigators per site-PI's guidance. Computer-based records will be maintained through the Veteran's Administration Computerized Patient Record System (CPRS), a secure network with password protection. A separate tracking database with participant identifiers that provide a link to the unique study IDs will be stored on a secure VA research server at each study site. Only deidentified data will be entered into the Redcap database by study personnel who are credentialed at the Birmingham VAMC through the research office.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will become available 1-year following the reporting of the primary and secondary outcome analyses.
Access Criteria: By study team permission

REFERENCES:
- [Derived] Markland AD, Goldstein KM, Beasley TM, Boyd EM, Zubkoff L, Kelly UA, Burgio KL, Vaughan CP. Remote Access to Urinary Incontinence Treatments for Women Veterans: The PRACTICAL Randomized Clinical Trial. JAMA Netw Open. 2025 Sep 2;8(9):e2532111. doi: 10.1001/jamanetworkopen.2025.32111. PMID 40956581
- [Derived] Hay-Smith EJC, Starzec-Proserpio M, Moller B, Aldabe D, Cacciari L, Pitangui ACR, Vesentini G, Woodley SJ, Dumoulin C, Frawley HC, Jorge CH, Morin M, Wallace SA, Weatherall M. Comparisons of approaches to pelvic floor muscle training for urinary incontinence in women. Cochrane Database Syst Rev. 2024 Dec 20;12(12):CD009508. doi: 10.1002/14651858.CD009508.pub2. PMID 39704322
- [Derived] Funada S, Yoshioka T, Luo Y, Sato A, Akamatsu S, Watanabe N. Bladder training for treating overactive bladder in adults. Cochrane Database Syst Rev. 2023 Oct 9;10(10):CD013571. doi: 10.1002/14651858.CD013571.pub2. PMID 37811598
- [Derived] Markland AD, Vaughan CP, Goldstein KM, Hastings SN, Kelly U, Beasley TM, Boyd EM, Zubkoff L, Burgio KL. Optimizing remote access to urinary incontinence treatments for women veterans (PRACTICAL): Study protocol for a pragmatic clinical trial comparing two virtual care options. Contemp Clin Trials. 2023 Oct;133:107328. doi: 10.1016/j.cct.2023.107328. Epub 2023 Sep 1. PMID 37659594

DOCUMENTS (1):
  • Informed Consent Form (2022-06-24): https://cdn.clinicaltrials.gov/large-docs/53/NCT04237753/ICF_000.pdf